CLINICAL TRIAL: NCT00994214
Title: Phase II, Open, Randomised, Parallel Group, Noncomparative Multicentre Study to Assess the Efficacy and Safety of Repeated Subcutaneous (S.C.) Administration of Different Doses of BIM 23A760 in Acromegalic Patients
Brief Title: Study to Assess the Efficacy and Safety of Repeated Administration of BIM 23A760 in Patients With Acromegaly
Acronym: TULIPIA
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Preliminary data from this study does not support expected inhibition of GH and IGF-1
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2-55-52060-003; 2009-010787-42 (EudraCT Number)
Record Dates: First submitted 2009-10-13; First posted 2009-10-14 (Estimated); Results first posted 2016-02-10 (Estimated); Last update posted 2019-11-22 (Actual); Status verified 2019-11

CONDITIONS: Acromegaly
MeSH Terms: conditions — Acromegaly | interventions — TBR-760

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- BIM 23A760 1 mg (Experimental)
  Interventions: Drug: BIM 23A760
- BIM 23A760 2 mg (Experimental)
  Interventions: Drug: BIM 23A760
- BIM 23A760 4 mg (Experimental)
  Interventions: Drug: BIM 23A760
- BIM 23A760 6 mg (Experimental)
  Interventions: Drug: BIM 23A760

INTERVENTIONS:
Drug: BIM 23A760 — Subcutaneous injections of BIM23A760 once a week. Until progression or unacceptable toxicity develops.

SUMMARY:
The purpose of this study is to assess the efficacy of repeated subcutaneous (under the skin) injections at different doses of BIM 23A760 on growth hormone and insulin-like growth factor-1 levels in patients with acromegaly after 6 months of treatment.

ELIGIBILITY:
Inclusion Criteria:

* IGF-1 ≥1.3 x upper limit normal (ULN)
* Nadir serum GH concentration ≥0.4 ng/mL in an oral glucose tolerance test (OGTT)
* Patient must have documentation supporting the diagnosis of acromegaly, including elevated GH and/or insulin-like growth factor-1 (IGF-1) levels.

Exclusion Criteria:

* The patient has received long acting somatostatin analogues within 6 months of study entry
* The patient has undergone radiotherapy at any time prior to study entry
* The time between pituitary surgery (if any) and study entry is less than 6 weeks
* The patient suffers from macroadenoma with visual field defects due to chiasmatic compression

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2009-10; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (23):
- United States (3):
  - Pituitary Center, Los Angeles, California
  - Massachusetts General Hospital / Neuroendocrine Unit, Boston, Massachusetts
  - Oregon University, Dept. of Endocrinology and Neurosurgery, Portland, Oregon
- Belgium (2):
  - UZ Leuven, Leuven
  - Centre Hospitalier Universitaire de Liège, Liège
- Brazil (2):
  - Hospital Universitário Clementino Fraga Filho, Rio de Janeiro
  - Hospital das Clínicas de São Paulo, São Paulo
- Czechia (2):
  - University Hospital Olomouc, Clinic of Internal Medicine, Olomouc
  - General University Hospital, Clinic of Internal Medicine,, Prague
- France (2):
  - Hôpital Bicêtre, Le Kremlin-Bicêtre
  - Hôpital de la Timone, Marseille
- P. Stradins Clinical University Hospital, Riga, Latvia
- Lithuania (2):
  - Kaunas Medical University Hospital, Kaunas
  - Vilnius University Hospital "Santariskiu Klinikos", Vilnius
- Mexico (2):
  - UIM Endocrinología Experimental, Hospital de Especialidades, Mexico City
  - Insituto Nacional de Neurologia y Neurocirugia, México
- Department of Endocrinology, Erasmus MC, Rotterdam, Netherlands
- Voivodeship Specialistic Hospital No 3, Rybnik, Poland
- "C.I. Parhon" National Institute of Endocrinology, Bucharest, Romania
- Karolinska University Hospital, Stockholm, Sweden
- Ukraine (3):
  - Academy of Medical Science of Ukraine, Department of Clinical Endocrinology, Kharkiv
  - Administration of Medical Services and Rehabilitation of "ARTEM", Kyiv
  - National Medical University n.a. M.I.Pirogov, Vinnitsa

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a multicentre study conducted at 36 investigational sites in 16 countries: Czech Republic, Lithuania, Poland, Romania, Ukraine, Latvia, USA, United Kingdom (UK), Italy, Mexico, Brazil, France, Belgium, Netherlands, Germany and Sweden.
Pre-assignment Details: Screened subjects were 109 and screen failures were 33. Subjects randomised and treated in part A were 76. Subjects completed part A were 21 and subjects entered Part B were 12, excluding 9 subjects, who chose not to continue in part B. No subjects completed the study.
Groups:
- Arm A: BIM 23A760 1 mg: BIM 23A760 1 mg subcutaneous 24 weekly injections.
- Arm B: BIM 23A760 2 mg: BIM 23A760 2 mg subcutaneous 24 weekly injections.
- Arm C: BIM 23A760 4 mg: BIM 23A760 4 mg subcutaneous 24 weekly injections.
- Arm D: BIM 23A760 6 mg: BIM 23A760 6 mg subcutaneous 24 weekly injections.
Period: ITT (Intention-to-Treat) - Part A
Arm/Group | Arm A: BIM 23A760 1 mg | Arm B: BIM 23A760 2 mg | Arm C: BIM 23A760 4 mg | Arm D: BIM 23A760 6 mg
Started | 19 | 19 | 18 | 20
Completed | 5 | 6 | 5 | 5
Not Completed | 14 | 13 | 13 | 15
Not completed — Adverse Event | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0
Not completed — Withdrawn - Study termination by sponsor | 13 | 12 | 13 | 14
Period: ITT (Intention-to-Treat) - Part B
Arm/Group | Arm A: BIM 23A760 1 mg | Arm B: BIM 23A760 2 mg | Arm C: BIM 23A760 4 mg | Arm D: BIM 23A760 6 mg
Started | 4 (1 subject did not enter Part B Arm A) | 3 (3 subjects did not enter Part B Arm B) | 2 (3 subjects did not enter Part B Arm C) | 3 (2 subjects did not enter Part B Arm D)
Received Maximum Dose of 1mg | 0 | 0 | 0 | 0
Received Maximum Dose of 2mg | 3 | 0 | 0 | 0
Received Maximum Dose of 4mg | 1 | 3 | 0 | 0
Received Maximum Dose of 6mg | 0 | 0 | 2 | 3
Completed | 0 | 0 | 0 | 0
Not Completed | 4 | 3 | 2 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1
Not completed — Withdrawn - Study termination by sponsor | 4 | 3 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: BIM 23A760 1 mg | Arm B: BIM 23A760 2 mg | Arm C: BIM 23A760 4 mg | Arm D: BIM 23A760 6 mg | Total
Number analyzed (Participants) | 19 | 19 | 18 | 20 | 76
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.8 (11.3) | 48.7 (11.2) | 40.3 (11.3) | 43.4 (12.9) | 43.8 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 13 | 6 | 13 | 42
  Male | 9 | 6 | 12 | 7 | 34
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian/White | 17 | 14 | 13 | 18 | 62
  Multiple race | 2 | 5 | 5 | 2 | 14
Region of Enrollment [Number; unit: Participants] — ITT population
  Participants
    Belgium | 1 | 1 | 0 | 0 | 2
    Brazil | 1 | 1 | 3 | 5 | 10
    Czech Republic | 1 | 1 | 0 | 1 | 3
    Lithuania | 1 | 1 | 3 | 1 | 6
    Mexico | 2 | 4 | 4 | 1 | 11
    Netherlands | 2 | 0 | 0 | 1 | 3
    Poland | 1 | 1 | 0 | 0 | 2
    Romania | 4 | 3 | 1 | 4 | 12
    Ukraine | 6 | 4 | 4 | 6 | 20
    France | 0 | 1 | 0 | 1 | 2
    United States | 0 | 2 | 1 | 0 | 3
    Latvia | 0 | 0 | 1 | 0 | 1
    Sweden | 0 | 0 | 1 | 0 | 1
Height [Mean (Standard Deviation); unit: cm] | 170.1 (8.1) | 170.3 (13.2) | 175.0 (10.1) | 166.4 (8.6) | 170.3 (10.4)
Diabetic status at entry [Number; unit: Participants]
  Diabetic | 2 | 1 | 2 | 2 | 7
  Non-diabetic | 17 | 18 | 16 | 18 | 69
Insulin-like growth factor 1 (IGF-1) [Median (Full Range); unit: Percentage of ULN(Upper limit of number)] | 307 [146 to 690] | 315 [176 to 508] | 382 [168 to 549] | 335 [157 to 539] | 333 [146 to 690]
Growth Hormone (GH) [Mean (Standard Deviation); unit: ng/mL] | 16.79 (24.56) | 20.99 (59.28) | 28.60 (64.83) | 26.59 (63.47) | 23.21 (55.54)
Baseline Prolactin [Mean (Standard Deviation); unit: μg/L]
  Males (n=A:9,B:6,C:12, D:7, and Total:34) | 11.506 (14.233) | 34.113 (49.588) | 41.657 (60.965) | 83.036 (131.024) | 40.86 (72.52)
  Pre-menopausal female(n=A:4,B:4,C:4,D:7,&Totl:19) | 19.838 (15.247) | 26.158 (19.798) | 35.608 (25.536) | 23.634 (23.778) | 25.88 (21.94)
  Post-menopausal female(n=A:6,B:9,C:2,D:6,&Totl:23) | 8.420 (3.167) | 16.409 (24.232) | 7.870 (0.693) | 25.118 (39.986) | 15.85 (25.89)
Ring Finger Circumference [Mean (Standard Deviation); unit: mm] | 70.2 (5.6) | 68.5 (6.2) | 71.2 (4.7) | 68.4 (6.3) | 69.53 (5.75)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Mean GH ≤2.5 ng/mL and Normalised IGF-1
Time Frame: At Month 6
Population: Intention-to-Treat (ITT) population: All randomized subjects who received at least one dose of study medication. N=Number of subjects attended Month 6 (visit 9).
Measure: Number; unit: Percentage of subjects
Arm/Group | Arm A: BIM 23A760 1 mg | Arm B: BIM 23A760 2 mg | Arm C: BIM 23A760 4 mg | Arm D: BIM 23A760 6 mg
Number analyzed (Participants) | 6 | 7 | 5 | 5
Percentage of subjects
  Mean GH ≤2.5 ng/mL and Normalised IGF-1: Yes | 0 | 0 | 0 | 0
  Mean GH ≤2.5 ng/mL and Normalised IGF-1: No | 83.3 | 100.0 | 100.0 | 100.0
  Missing | 16.7 | 0 | 0 | 0

2. Secondary Outcome: Percentage of Subjects With Mean GH ≤2.5 ng/mL and Normalised IGF-1
Time Frame: At Month 3
Population: ITT population. N=Number of subjects attended Month 3 (visit 7).
Measure: Number; unit: Percentage of subjects
Arm/Group | Arm A: BIM 23A760 1 mg | Arm B: BIM 23A760 2 mg | Arm C: BIM 23A760 4 mg | Arm D: BIM 23A760 6 mg
Number analyzed (Participants) | 12 | 13 | 12 | 13
Percentage of subjects
  Mean GH ≤2.5 ng/mL and Normalised IGF-1: Yes | 0 | 0 | 0 | 7.7
  Mean GH ≤2.5 ng/mL and Normalised IGF-1: No | 100 | 100 | 100 | 92.3
  Missing | 0 | 0 | 0 | 0

3. Secondary Outcome: Percentage of Subjects With Mean GH ≤2.5 ng/mL and Normalised IGF-1
Time Frame: At Month 1
Population: ITT population. N=Number of subjects attended Month 1 (visit 5).
Measure: Number; unit: Percentage of subjects
Arm/Group | Arm A: BIM 23A760 1 mg | Arm B: BIM 23A760 2 mg | Arm C: BIM 23A760 4 mg | Arm D: BIM 23A760 6 mg
Number analyzed (Participants) | 19 | 18 | 18 | 20
Percentage of subjects
  Mean GH ≤2.5 ng/mL and Normalised IGF-1: Yes | 5.3 | 0 | 0 | 5.0
  Mean GH ≤2.5 ng/mL and Normalised IGF-1: No | 94.7 | 100 | 100 | 95.0
  Missing | 0 | 0 | 0 | 0

4. Secondary Outcome: Percent Change From Baseline in the Mean GH From 0-3 Hours at Months 1, 3 and 6
Description: Percentage change from Baseline at month X = (Mean GH at month X - Mean GH at baseline) x 100 / Mean GH at baseline
Time Frame: 0-3 hr on Baseline (Day 1) and Months 1, 3 and 6
Population: N=Number of patients randomised to treatment in IGF-1 <2.5 x upper limit of normal (ULN) stratum and IGF-1 ≥2.5 x ULN stratum.
Measure: Mean (Standard Deviation); unit: Percentage of change in mean GH
Arm/Group | Arm A: BIM 23A760 1 mg | Arm B: BIM 23A760 2 mg | Arm C: BIM 23A760 4 mg | Arm D: BIM 23A760 6 mg
Number analyzed (Participants) | 15 | 15 | 15 | 16
Percentage of change in mean GH
  At Month 1: IGF-1<2.5 x ULN | 4.10 (53.03) | -0.55 (23.98) | -9.92 (71.51) | -17.59 (41.82)
  At Month 3: IGF-1<2.5 x ULN | 29.26 (45.97) | -18.99 (21.36) | 17.48 (127.97) | -28.84 (43.25)
  At Month 6: IGF-1<2.5 x ULN | 71.44 (35.97) | 3.32 (9.09) | 82.45 (0) | -38.21 (27.27)
  At Month 1: IGF-1≥2.5 x UL | -39.20 (30.33) | -22.24 (34.72) | -10.64 (51.18) | -23.63 (39.57)
  At Month 3: IGF-1≥2.5 x UL | -26.14 (39.60) | -22.35 (31.71) | -7.64 (30.11) | -20.53 (42.23)
  At Month 6: IGF-1≥2.5 x UL | -36.15 (45.63) | 15.28 (82.56) | -10.43 (28.90) | -19.47 (68.90)

5. Secondary Outcome: Changes in IGF-1
Time Frame: Baseline (Day 1) and Month 6
Population: ITT population
Measure: Mean (Standard Deviation); unit: Percentage of ULN
Arm/Group | Arm A: BIM 23A760 1 mg | Arm B: BIM 23A760 2 mg | Arm C: BIM 23A760 4 mg | Arm D: BIM 23A760 6 mg
Number analyzed (Participants) | 19 | 19 | 18 | 20
Percentage of ULN | -51.30 (136.66) | -53.31 (80.57) | -40.53 (56.65) | -85.91 (95.34)

6. Secondary Outcome: Percentage Change in Ring Finger Circumference
Description: Percentage change from Baseline at month X = (Ring finger circumference at month X - ring finger circumference at baseline) x 100 / ring finger circumference at baseline.
Time Frame: Baseline (Day 1) and Month 6
Population: ITT population. N=Number of subjects attended Month 6 (visit 9).
Measure: Mean (Standard Deviation); unit: Percentage of Change in Ring Finger circ
Arm/Group | Arm A: BIM 23A760 1 mg | Arm B: BIM 23A760 2 mg | Arm C: BIM 23A760 4 mg | Arm D: BIM 23A760 6 mg
Number analyzed (Participants) | 6 | 7 | 5 | 5
Percentage of Change in Ring Finger circ | -3.518 (3.688) | -1.469 (2.120) | -0.678 (2.409) | -4.003 (3.367)

7. Secondary Outcome: Number of Subjects Reported Adverse Events During the Study
Description: For summaries of intensity and causality, individual patients may be reported in more than one category. In the event of multiple episodes of AEs being reported by the same patient during the study, the maximum intensity (severe > moderate > mild) and the most serious causality (related > not related) have been chosen.
  TEAE (Treatment emergent adverse event) are reported by Maximum Dose Received in Each Part of the Study.
Time Frame: Up to Visit 10 (An average of 6.5 Months)
Population: Safety Population
  Part B: Arm A: BIM 23A760 1 mg- 4 subjects from part B, Arm A were considered under other arms of part B based on the maximum dose received.
Measure: Number; unit: Participants
Arm/Group | Part A: Arm A: BIM 23A760 1 mg | Part A: Arm B: BIM 23A760 2 mg | Part A: Arm C: BIM 23A760 4 mg | Part A: Arm D: BIM 23A760 6 mg | Overall - Part A | Part B: Arm B: BIM 23A760 2 mg | Part B: Arm C: BIM 23A760 4 mg | Part B: Arm D: BIM 23A760 6 mg | Overall - Part B
Number analyzed (Participants) | 19 | 19 | 18 | 20 | 76 | 3 | 4 | 5 | 12
Participants
  Severe | 0 | 1 | 1 | 2 | 4 | 0 | 0 | 0 | 0
  Moderate | 3 | 8 | 4 | 7 | 22 | 0 | 0 | 3 | 3
  Mild | 11 | 9 | 12 | 15 | 47 | 0 | 1 | 1 | 2
  Related | 7 | 8 | 10 | 11 | 36 | 0 | 0 | 1 | 1
  Not Related | 8 | 9 | 6 | 11 | 34 | 0 | 1 | 3 | 4

ADVERSE EVENTS:
Time Frame: Up to Visit 10 (An average of 6.5 Months)
Description: Included Serious Adverse Events (SAEs) and Adverse Events (AEs) during treatment phase for Safety Population
  TEAE are reported by Maximum Dose Received in Each Part of the Study.
  4 subjects from part B, Arm A were considered under other arms of part B based on the maximum dose received.
Arm/Group | Part A: Arm A: BIM 23A760 1 mg | Part A: Arm B: BIM 23A760 2 mg | Part A: Arm C: BIM 23A760 4 mg | Part A: Arm D: BIM 23A760 6 mg | Overall - Part A | Part B: Arm B: BIM 23A760 2 mg | Part B: Arm C: BIM 23A760 4 mg | Part B: Arm D: BIM 23A760 6 mg | Overall - Part B
Serious Adverse Events (participants affected / at risk) | 1/19 | 2/19 | 0/18 | 0/20 | 3/76 | 0/3 | 0/4 | 2/5 | 2/12
Other Adverse Events (participants affected / at risk) | 11/19 | 12/19 | 12/18 | 15/20 | 50/76 | 0/3 | 1/4 | 4/5 | 5/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: Arm A: BIM 23A760 1 mg (N=19) | Part A: Arm B: BIM 23A760 2 mg (N=19) | Part A: Arm C: BIM 23A760 4 mg (N=18) | Part A: Arm D: BIM 23A760 6 mg (N=20) | Overall - Part A (N=76) | Part B: Arm B: BIM 23A760 2 mg (N=3) | Part B: Arm C: BIM 23A760 4 mg (N=4) | Part B: Arm D: BIM 23A760 6 mg (N=5) | Overall - Part B (N=12)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: Arm A: BIM 23A760 1 mg (N=19) | Part A: Arm B: BIM 23A760 2 mg (N=19) | Part A: Arm C: BIM 23A760 4 mg (N=18) | Part A: Arm D: BIM 23A760 6 mg (N=20) | Overall - Part A (N=76) | Part B: Arm B: BIM 23A760 2 mg (N=3) | Part B: Arm C: BIM 23A760 4 mg (N=4) | Part B: Arm D: BIM 23A760 6 mg (N=5) | Overall - Part B (N=12)
ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PANCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VERTIGO (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPOTHYROIDISM (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
EYE IRRITATION (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LACRIMATION INCREASED (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1) | 1 (2) | 1 (1) | 3 (5) | 6 (9) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 2 (3) | 1 (1) | 1 (10) | 2 (7) | 6 (21) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FLATULENCE (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GASTROINTESTINAL PAIN (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 2 (2) | 2 (3) | 2 (3) | 2 (5) | 8 (13) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PROCTALGIA (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VOMITING (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ADMINISTRATION SITE REACTION (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (7) | 1 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
APPLICATION SITE ERYTHEMA (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
APPLICATION SITE INDURATION (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ASTHENIA (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FATIGUE (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERTHERMIA (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INJECTION SITE ERYTHEMA (General disorders) | 0 (0) | 2 (4) | 1 (15) | 3 (10) | 6 (29) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INJECTION SITE INDURATION (General disorders) | 2 (2) | 2 (4) | 4 (5) | 1 (2) | 9 (13) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INJECTION SITE INFLAMMATION (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INJECTION SITE NODULE (General disorders) | 1 (1) | 1 (1) | 2 (4) | 2 (6) | 6 (12) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INJECTION SITE PAIN (General disorders) | 0 (0) | 0 (0) | 2 (6) | 2 (5) | 4 (11) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INJECTION SITE PRURITUS (General disorders) | 0 (0) | 2 (4) | 3 (16) | 3 (7) | 8 (27) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INJECTION SITE RASH (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INJECTION SITE REACTION (General disorders) | 0 (0) | 2 (4) | 0 (0) | 2 (9) | 4 (13) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INJECTION SITE SWELLING (General disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OEDEMA PERIPHERAL (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CYSTITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FUNGAL SKIN INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NASOPHARYNGITIS (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SINUSITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CONCUSSION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
WOUND (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLOOD AMYLASE INCREASED (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLOOD GLUCOSE INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLOOD PRESSURE DECREASED (Investigations) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLOOD PRESSURE DIASTOLIC INCREASED (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLOOD THYROID STIMULATING HORMONE DECREASED (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RED BLOOD CELLS URINE POSITIVE (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TRI-IODOTHYRONINE FREE INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
WHITE BLOOD CELLS URINE POSITIVE (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERCHOLESTEROLAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
IMPAIRED FASTING GLUCOSE (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RHEUMATOID ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SYNOVITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ACOUSTIC NEURITIS (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CARPAL TUNNEL SYNDROME (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DIZZINESS (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (2) | 5 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HEADACHE (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 3 (4) | 4 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPOAESTHESIA (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PARAESTHESIA (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PRESYNCOPE (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SYNCOPE (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TRIGEMINAL NEURALGIA (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INSOMNIA (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
POLLAKIURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MENSTRUATION DELAYED (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RESPIRATORY DISORDER (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERKERATOSIS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PRURITUS (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPOTENSION (Vascular disorders) | 0 (0) | 1 (1) | 3 (4) | 0 (0) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PERIPHERAL COLDNESS (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PHLEBITIS (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GASTRITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
CHOLELITHIASIS (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
CYTOLYTIC HEPATITIS (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
BLOOD PRESSURE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was terminated prematurely due to lack of efficacy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No